CLINICAL TRIAL: NCT06756373
Title: Adherence to International Guidelines Directed Risk Stratification and Management of Acute Pulmonary Embolism, an Egyptian Experience
Brief Title: Mangement of Pulmonary Emboli
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rania Abdelmoaz Farghaly, resident doctor, Assiut University
Other Study IDs: mangement of pulmonary emboli
Record Dates: First submitted 2024-12-17; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Pulmonary Embolism (Diagnosis)
Keywords: simplified pulmonary embolism l index; POPE
MeSH Terms: conditions — Pulmonary Embolism; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- To assess to which extent we are adherent to ESC guidelines 2019 in management of patients presented: Comparing ESC 2019 criteria for risk stratification and mortality with new scores [BOVA , modified FAST, PEITHO-3 models & POPE].
  -Comparing management and outcomes of in hospital and 30 days follow up of pulmonary embolism before and after starting PERT in our center

SUMMARY:
To assess to which extent we are adherent to ESC guidelines 2019 in management of patients presented with acute pulmonary embolism

DETAILED DESCRIPTION:
Pulmonary embolism (PE) is the third most frequent cardiovascular disease and is associated with a high mortality burden PE is defined as the obstruction of a pulmonary artery, mostly resulting from the dislodgement of thrombotic material from the lower limbs. It has a wide variety of presentations, ranging from an asymptomatic incidental finding to circulatory collapse and sudden death Pulmonary embolism response teams (PERTs) have emerged as a multidisciplinary team for managing acute pulmonary embolism, with a rapid activation process for multimodality assessment, risk stratification and best management especially for complex challenge cases. PERTs help in improving time to PE diagnosis; shorter time to initiation of anticoagulation reducing hospital length of stay, increasing use of advanced therapies as catheter directed therapies without an increase in bleeding complications with decreasing mortality

ELIGIBILITY:
Inclusion Criteria:

* No includion criteria

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: treatment of patient with pulmonary embolism according to ECS Guidlines
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2026-12-17 (Estimated); Study Completion 2027-12-17 (Estimated)

PRIMARY OUTCOMES:
mortality rate | 30 day
  mortality rate of pulmonary embolism

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gerardo F, Faria D, Silverio Antonio P, Baltazar Ferreira J, Beringuilho M, Ferreira H, Fialho I, Miranda I, Sa Pereira Y, Nunes-Ferreira A, Roque D, Santos MB, Morais C, Bravo Baptista S, Augusto JB. PrOgnosis in Pulmonary Embolism (PoPE): 30-Day mortality risk score based on five admission parameters. Rev Port Cardiol. 2024 Jan;43(1):1-8. doi: 10.1016/j.repc.2023.04.011. Epub 2023 Jul 7. English, Portuguese. PMID 37423312
- [Background] Leidi A, Bex S, Righini M, Berner A, Grosgurin O, Marti C. Risk Stratification in Patients with Acute Pulmonary Embolism: Current Evidence and Perspectives. J Clin Med. 2022 Apr 30;11(9):2533. doi: 10.3390/jcm11092533. PMID 35566658
- [Background] Cohen AT, Agnelli G, Anderson FA, Arcelus JI, Bergqvist D, Brecht JG, Greer IA, Heit JA, Hutchinson JL, Kakkar AK, Mottier D, Oger E, Samama MM, Spannagl M; VTE Impact Assessment Group in Europe (VITAE). Venous thromboembolism (VTE) in Europe. The number of VTE events and associated morbidity and mortality. Thromb Haemost. 2007 Oct;98(4):756-64. doi: 10.1160/TH07-03-0212. PMID 17938798
- [Background] ISTH Steering Committee for World Thrombosis Day. Thrombosis: a major contributor to the global disease burden. J Thromb Haemost. 2014 Oct;12(10):1580-90. doi: 10.1111/jth.12698. PMID 25302663